CLINICAL TRIAL: NCT03514771
Title: Early Non-Ablative Fractional Laser Resurfacing for Acne Scars After Treatment With Oral Isotretinoin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Smart (Other)
Responsible Party: Sponsor-Investigator, David Smart, Principal Investigator, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB_00087490
Record Dates: First submitted 2017-12-06; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic
MeSH Terms: conditions — Hypertrophy | interventions — Isotretinoin; Valacyclovir

STUDY DESIGN:
Intervention Model Description: All subjects will have one side of the face (Right-Left) treated with the laser and the other side will be untreated to act as a control.
Who Masked: Outcomes Assessor
Masking Description: Efficacy evaluations of photographs will be performed by two trained and experienced evaluators who are blinded to which side of the face has been treated, and which side of the face has not been treated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Subjects (Other): All subjects will have one side of their face treated with the laser and one side not treated to serve as the control.
  Interventions: Device: Fraxel DUAL 1550/1927; Drug: oral isotretinoin; Drug: oral valacyclovir

INTERVENTIONS:
Device: Fraxel DUAL 1550/1927
Drug: oral isotretinoin — oral isotretinoin
Drug: oral valacyclovir — Oral valacyclovir

SUMMARY:
Patients who have completed have completed a cumulative dose of >=120miligram/kilogram oral isotretinoin within the last 30 days, and has mild to moderate acne scarring will be randomized, into a right-left comparison study using Fraxel DUAL (Solta Medical) laser on one side of the face, and no treatment on the other side of the face. Subejcts will receive treatments at week 0, week 4, and week 8. Photographs will be taken after each treatment, 7 days after each treatment, and 4 months after last treatment. Photographs will be reviewed by blind assessors who will analyze the pre- and post-treatment photographs to measure change.

DETAILED DESCRIPTION:
Approximately 15 patients who are over 18 years or older, have completed a cumulative dose of >=120miligram/kilogram oral isotretinoin within the last 30 days, and has mild to moderate acne scarring will be randomized, into a right-left comparison study.

One side of the face will be randomized to NAFR treatment and other side to control (no treatment) using a random number generator. Subjects will apply topical anesthetic (Benzocaine / Lidocaine / Tetracaine 20% / 8% / 4% Ointment) to the entire face one hour prior to treatment. The NAFR operator will be notified of which side is to be treated with NAFR.

To ensure blinded evaluations, the same unblinded investigator will perform all the laser treatments, whereas efficacy evaluations will be performed by two trained and experienced evaluators who are blinded to the treatment assignment. Evaluations for adverse effects will be carried out by the unblinded NAFR (during and immediately post treatment) and the two blinded investigators at prescribed intervals.

Treatments:

Laser procedure will be performed to the entire assigned half of the face with Fraxel DUAL (Solta Medical) with the following settings: 1550 nanometer; 35 to 40 millijoules/microthermal zone, treatment level from 7 to 10, corresponding to treatment coverage of 20% to 35%. The treatment protocol was modified slightly depending on the individual scar characteristics (depth, width, and type).

The patients will receive a total of three laser treatments using NAFR. Successive treatments will be separated by 1 month. During all treatments, pain will be assessed as ''mild, moderate, or severe.'' Post-treatment instructions will include the use of a mild soap, sunscreen in the morning, and a non-comedogenic moisturizing cream in the evening twice daily for three days. Oral valacyclovir (1 gram daily) will be prescribed for patients for prophylaxis of herpetic infection.

Evaluations:

Photographic documentation using identical camera settings, lighting, and patient positioning will be obtained at baseline, before each treatment session, 7-days after each session, and 4 months after the final treatment.

Primary Efficacy Measure:

Wound healing will be assessed after 7 days of each treatment and at the end of the study (4 month after last treatment) in all patients. This will be performed by 2 blinded evaluators who will analyze the pre and post-treatment photographs.

Secondary Efficacy Measure:

Secondary study endpoints will be improvement of acne scarring, assessment of treatment tolerability (adverse effects, pain assessment, and patient satisfaction and preference.

Improvement in acne scarring will be graded by two independent blinded physicians using a quartile grading scale (1 = 1% to 25%, 2 =26% to 50%, 3 =51% to 75%, 4 = >76%). All grading physicians will be blinded to the total number of treatments and which photographs were baseline and follow-up at 4 month after last treatment.

Evaluations for immediate and delayed adverse effects of the treatments, including erythema, edema, blistering, crusting, scarring, and hyperpigmentation, graded on a 4-point scale (0 = absent, 1= mild, 2 = moderate, and 3 = severe) will be carried out at each visit.

Patients will also assess the intensity of pain post-treatment using a visual analogue scale (VAS) (0 = absence of pain, 10 = most-severe pain).

Patient assessment of efficacy would be reflected by their judgment of which side of the face responded best to treatment. Patient preference can then be assessed at the end of the study asking, "would you recommend NAFR treatment for acne scarring to others?"

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Completed cumulative dose of >=120 miligram/kilogram oral isotretinoin within the last 30 days
* Mild-moderate acne scarring of all types (icepick, boxcar, rolling)

Exclusion Criteria:

* Pregnant or nursing women
* History of porphyria, allergy to porphyrins, or photodermatosis
* Active infectious disease
* Severe acne scarring
* Propensity to hypertrophic or keloid scarring
* Immunosuppression
* Laser or any cosmetic treatment in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
The adverse events associated with early non-ablative fractional laser resurfacing (NAFR) for mild-moderate acne scars after treatment with oral isotretinoin compared to control (non-treated side of the face). | Baseline visit through 4 month follow-up
  Adverse Events

SECONDARY OUTCOMES:
To evaluate the efficacy of early non-ablative fractional laser resurfacing (NAFR) for mild-moderate acne scars after treatment with oral isotretinoin compared to control (non-treated side of the face). | up to 4-months follow up
  To compare acne improvement using a quartile grading scale (1 = 1% to 25%, 2 =26% to 50%, 3 =51% to 75%, 4 = >76%). improvement). Photos taken at each treatment.

IPD SHARING:
Plan to Share IPD: No